CLINICAL TRIAL: NCT00768274
Title: A Safety, Pharmacokinetic, and Pharmacodynamic Assessment of 28-Day Oral Dosing of RVX000222 in Healthy Subjects and Subjects With Low High Density Lipoprotein (HDL)
Brief Title: Safety, Pharmacokinetic Study of RVX000222 in Healthy Subjects and Subjects With Low HDL Cholesterol
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Resverlogix Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RVX222-CS-003
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2016-07

CONDITIONS: Dyslipidemia; Atherosclerosis; Acute Coronary Syndrome; Cardiovascular Disease
Keywords: Cholesterol; High density lipoprotein; Dyslipidemia; Atherosclerosis; Apolipoprotein A-I
MeSH Terms: conditions — Dyslipidemias; Atherosclerosis; Acute Coronary Syndrome; Cardiovascular Diseases | interventions — apabetalone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Arm A (Experimental): Low-dose apabetalone (RVX000222) or placebo
  Interventions: Drug: RVX000222; Drug: Placebo
- Arm B (Experimental): apabetalone (RVX000222) Dose-escalation or placebo
  Interventions: Drug: RVX000222; Drug: Placebo
- Arm C (Experimental): high-dose apabetalone (RVX000222) or placebo
  Interventions: Drug: RVX000222; Drug: Placebo

INTERVENTIONS:
Drug: RVX000222 — RVX000222 twice daily (b.i.d.) for 28 days
  Other Names: RVX-208; apabetalone
Drug: Placebo — Placebo twice daily (b.i.d.) for 28 days

SUMMARY:
The purpose of this study is to investigate an oral formulation of RVX000222 for safety, pharmacokinetic and efficacy in healthy subjects.

DETAILED DESCRIPTION:
One-third of the US population, almost 80 million adults, have cardiovascular disease and mortality associated with heart disease which still remains a leading cause of death around the world. The major risk factors for cardiovascular disease associated with atherosclerosis is dyslipidemia, characterized by high levels of low density lipoprotein (LDL) and/or low levels of high density lipoprotein (HDL).

HDL has a well established role in atherosclerosis and cardiovascular disease protection. HDL mediates the removal of cholesterol from the atherosclerotic plaques for elimination from the body. The major component of HDL consists of apolipoprotein A-I (ApoA I). Recent intervention studies with synthetic HDL particles and recombinant ApoA-I have shown that HDL has the capacity to reverse coronary atherosclerosis.

RVX000222 is a member of a novel class of small molecules that are candidates for the treatment of dyslipidemia by increasing plasma levels of ApoA-I and HDL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the following criteria may be enrolled:

  1. Be men or women between 18 and 65 years old, inclusive
  2. Weigh between 60 kg and 110 kg, inclusive, and have a BMI ≥25 kg/m2.
  3. Healthy volunteers with normal or low HDL
  4. If female, non-pregnant (as determined by a negative serum pregnancy test at Screening), non-lactating, and not of childbearing-potential or willing to practice an acceptable form of birth control. If male, be willing to practice an acceptable form of birth control.

Exclusion Criteria:

* Subjects who meet any of the following criteria will not be enrolled:

  1. Have presently, or have a history of, clinically significant disease, including cardiovascular, gastrointestinal, renal, hepatic, pulmonary, endocrine, hematologic, vascular, immunologic, metabolic, neurological, or collagen disease, as judged by the Investigator.
  2. Have active cholecystitis or gallbladder symptoms within 60 days prior to Check-in (subjects who have had a cholecystectomy are not excluded from this study).
  3. Have had a clinically significant illness, in the opinion of the Investigator, within 30 days prior to Check-in.
  4. Have hypertension that is currently being treated, or uncontrolled hypertension
  5. Have a serum creatinine >1.5 mg/dL, hemoglobin <11.2 g/dL, or white blood cell count <4000/μL.
  6. Have positive test results for HIV, hepatitis A, B, or C.
  7. Have a positive result on drug screen testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety, pharmacokinetics and changes in lipid parameters from baseline and placebo. | 1-month

CONTACTS AND LOCATIONS:
Overall Officials: Allan Gordon, MD, PhD, Study Director — Resverlogix Corp
Locations (1):
- Covance Clinical Research Unit, Inc., Dallas, Texas, United States